CLINICAL TRIAL: NCT05923411
Title: A PHASE 1, RANDOMIZED, OPEN-LABEL, PARALLEL-GROUP, SINGLE-DOSE STUDY IN HEALTHY PARTICIPANTS TO INVESTIGATE THE RELATIVE BIOAVAILABILITY OF TWO TABLET FORMULATIONS OF PF-07220060, AND TO INVESTIGATE THE EFFECT OF FOOD AND A PROTON PUMP INHIBITOR ON THE RELATIVE BIOAVAILABILITY OF PF-07220060
Brief Title: A Study for Multiple Tablet Forms of The Study Medicine (PF-07220060) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C4391007
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Healthy Participants
Keywords: Food-effect; Relative Bioavailability; Pharmacokinetics; Proton Pump Inhibitor (PPI); Cyclin-Dependent Kinase 4 (CDK4) inhibitor; Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1 (Experimental): Participants will receive PF-07220060 tablet by mouth
  Interventions: Drug: Single dose of PF-07220060 as first Tablet Formulation
- Cohort 2 (Experimental): Participants will receive PF-07220060 tablet by mouth
  Interventions: Drug: Single dose of PF-07220060 as second Tablet Formulation
- Cohort 3 (Experimental): Participants will receive PF-07220060 tablet by mouth
  Interventions: Drug: Single dose of PF-07220060 as first Tablet Formulation
- Cohort 4 (Experimental): Participants will receive PF-07220060 tablet by mouth
  Interventions: Drug: Single dose of PF-07220060 as second Tablet Formulation
- Cohort 5 (Experimental): Participants will receive PF-07220060 tablet by mouth
  Interventions: Drug: Single dose of PF-07220060 as a Tablet Formulation
- Cohort 6 (Experimental): Participants will receive PF-07220060 and Rabeprazole tablets by mouth
  Interventions: Drug: Single dose of PF-07220060 as a Tablet formulation under Rabeprazole administration
- Cohort 7 (Experimental): Participants will receive PF-07220060 and Rabeprazole tablet by mouth
  Interventions: Drug: Single dose of PF-07220060 as a Tablet formulation under Rabeprazole administration
- Cohort 8 (Experimental): Participants will receive PF-07220060 tablet by mouth
  Interventions: Drug: Single dose of PF-07220060 as third tablet formulation

INTERVENTIONS:
Drug: Single dose of PF-07220060 as first Tablet Formulation — A single dose of PF-07220060 as the first Tablet Formulation administered under fasting conditions.
  Other Names: Cohort 1, first Tablet Formulation, Fasted
  Arms: Cohort 1
Drug: Single dose of PF-07220060 as second Tablet Formulation — A single dose of PF-0720060 as the second Tablet Formulation administered under fasting conditions
  Other Names: Cohort 2, second Tablet Formulation, Fasted
  Arms: Cohort 2
Drug: Single dose of PF-07220060 as first Tablet Formulation — A single dose of PF-07220060 as the first Tablet Formulation administered under fasting conditions at a second dose level
  Other Names: Cohort 3, first Tablet Formulation, Second Dose Level, Fasted
  Arms: Cohort 3
Drug: Single dose of PF-07220060 as second Tablet Formulation — A single dose of PF-07220060 as the second Tablet Formulation administered under fasting conditions at a second dose level
  Other Names: Cohort 4, second Tablet Formulation, Second Dose level, Fasted
  Arms: Cohort 4
Drug: Single dose of PF-07220060 as a Tablet Formulation — A single dose of PF-07220060 as a tablet formulation administered under fed conditions
  Other Names: Cohort 5, Fed
  Arms: Cohort 5
Drug: Single dose of PF-07220060 as a Tablet formulation under Rabeprazole administration — A 2-treatment fixed sequence of single dose of PF-07220060 tablets under fasting conditions followed by a single dose of PF-07220060 tablets under Proton Pump Inhibitor (PPI) administration under fasting condition (following a 7 day oral rabeprazole tablets daily administration).
  Other Names: Cohort 6, Fasted PPI
  Arms: Cohort 6
Drug: Single dose of PF-07220060 as a Tablet formulation under Rabeprazole administration — A 2-treatment fixed sequence of a single dose of PF-07220060 tablet given with moderate-fat, standard-calorie meal followed by a single dose of PF-07220060 tablet given with moderate-fat, standard-calorie meal and under PPI administration (following a 7 day oral rabeprazole tablets daily administration)
  Other Names: Cohort 7, Fed PPI
  Arms: Cohort 7
Drug: Single dose of PF-07220060 as third tablet formulation — A 2-period randomized 2-sequence cross over of a single dose of PF-07220060 as first and third tablet formulation under fasting conditions with a 6-day washout in between them
  Other Names: Cohort 8, third tablet formulation
  Arms: Cohort 8

SUMMARY:
The purpose of this study is to compare multiple formulations of PF-07220060 in terms of their uptake into the blood stream. The study will assess the effects of food and Rabeprazole on the uptake of PF-07220060. Rabeprazole belongs to a type of medications called proton pump inhibitors. In reality, some patients may take both PF-07220060 and rabeprazole together.

This study is seeking participants that are:

- Healthy male or female aged 18 to 65 years

Participants in this study will receive PF-07220060 once or twice by mouth. The participants may receive different tablets for PF-07220060. Some participants will take a meal before receiving PF-07220060. In addition, some participants will take rabeprazole by mouth for 7 days before taking PF-07220060.

The study will compare experiences of people receiving different formulations of PF-07220060. Experiences of people taking food and rabeprazole with PF-07220060 will be compared to those on PF-07220060 alone. This will help understand how much PF-07220060 is taken up into the blood. It will also help understand how meal and Rabeprazole medicine changes the uptake of PF-07220060 into the blood.

Participants will take part in the study for a maximum of 74 days. During this time, they will have to stay onsite for 5 to 13 days. There will be up to 2 onsite study visits.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring
* BMI of 17.5-30.5 kg/m2; and a total body weight >50 kg (110 lb).
* Evidence of a personally signed and dated ICD indicating that the participant has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
* History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg), or hepatitis B surface antigen (HCVAb). Hepatitis B vaccination is allowed.
* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

Prior/Concomitant Therapy:

* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention.
* Previous exposure to PF-07220060 or participation in studies requiring PF-07220060 administration.
* A positive urine drug test/urine cotinine test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2023-07-11 (Actual); Primary Completion 2024-06-23 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time(AUCinf) of PF-07220060 to estimate relative bioavailability of PF-07220060 two tablet formulations | 0 (pre-dose), 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours PF-07220060 post-dose
Maximum Observed Plasma Concentration (Cmax) of PF-07220060 to estimate relative bioavailability of PF-07220060 two tablet formulations | 0 (pre-dose), 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours PF-07220060 post-dose

SECONDARY OUTCOMES:
AUCinf of PF-07220060 to estimate relative bioavailability of PF-07220060 two tablet formulations at a second dose level | 0 (pre-dose), 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours PF-07220060 post-dose
Cmax of PF-07220060 to estimate relative bioavailability of PF-07220060 two tablet formulations at a second dose level | 0 (pre-dose), 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours PF-07220060 post-dose
Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time(AUCinf) of PF-07220060 to estimate relative bioavailability of PF-07220060 two tablet formulations (third formulation) | 0 (pre-dose), 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, and 96 hours PF-07220060 post-dose
Maximum Observed Plasma Concentration (Cmax) of PF-07220060 to estimate relative bioavailability of PF-07220060 two tablet formulations (third formulation) | 0 (pre-dose), 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, and 96 hours PF-07220060 post-dose
AUCinf of PF-07220060 to estimate the effect of a high-fat, high-calorie meal on the bioavailability of a PF-07220060 tablet formulation | 0 (pre-dose), 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours PF-07220060 post-dose
Cmax of PF-07220060 to estimate the effect of a high-fat, high-calorie meal on the bioavailability of a PF-07220060 tablet formulation | 0 (pre-dose), 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours PF-07220060 post-dose
AUCinf of PF-07220060 to estimate the effect of a PPI (rabeprazole) on the bioavailability of a PF-07220060 tablet formulation under fasted condition | 0 (pre-dose), 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours PF-07220060 post-dose
Cmax of PF-07220060 to estimate the effect of a PPI (rabeprazole) on the bioavailability of a PF-07220060 tablet formulation under fasted condition | 0 (pre-dose), 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours PF-07220060 post-dose
AUCinf of PF-07220060 to estimate the effect of a PPI (rabeprazole) on the bioavailability of a PF-07220060 tablet formulation under fed condition | 0 (pre-dose), 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours PF-07220060 post-dose
Cmax of PF-07220060 to estimate the effect of a PPI (rabeprazole) on the bioavailability of a PF-07220060 tablet formulation under fed condition | 0 (pre-dose), 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours PF-07220060 post-dose
Number of Participants With Laboratory Abnormalities | From baseline up to 28 days after PF-07220060 dose
Number of Participants With Clinically Significant Change in Electrocardiogram (ECG) Findings | From baseline up to 28 days after PF-07220060
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | From baseline up to 28 days after PF-07220060
Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs) | From baseline up to 28 days after PF-07220060 dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4391007